CLINICAL TRIAL: NCT06206759
Title: Vitamin C Administration and Triglycerides Level in Critical Care Patients: a Retrospective Study
Brief Title: Vitamin C Administration and Triglycerides Level in Critical Care Patients
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0318-23-MMC
Record Dates: First submitted 2023-12-19; First posted 2024-01-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group- ICU patients treated with vitamin C: ICU patients treated with vitamin C
  Interventions: Drug: administration of vitamin C
- control group- ICU patients not treated with vitamin C: ICU patients not treated with vitamin C

INTERVENTIONS:
Drug: administration of vitamin C — administration of vitamin C to ICU patients
  Groups: study group- ICU patients treated with vitamin C

SUMMARY:
Vitamin C (ascorbic acid) is a water-soluble vitamin with antioxidant properties. Previous studies showed that the administration of vitamin C was associated with decreased triglyceride (TG) levels in ambulatory patients, especially in patients with type 2 diabetes. The decrease in TG level was more significant the younger the patient's age (less than 52.8 years), the longer the administration of vitamin C lasted (over 12 weeks) and the higher the daily dose was (over 1 gram per day) (2). However, we did not find any studies that examined the relationship between administration of vitamin C and lowering of TG level in critical patients in intensive care. High TG levels are often found in these patients, secondary to sepsis, administration of propofol by continuous infusion, administration of TPN, pancreatitis, liver failure and chronic dyslipidemia, diabetes and chronic renal failure. High TG levels in these patients may cause pancreatitis secondary to elevated TG, and we take several actions to lower TG levels in the unit when they exceed 500 mg per dL in order to avoid these complications. The actions taken include starting treatment with fibrates and/or statins, giving high-dose insulin, stopping the propofol drip and changing it to another hypnotic drug (usually midazolam), and giving fat-free TPN instead of fat-containing TPN. There are of course disadvantages to these interventions, such as drug interactions, longer clearance time and higher incidence of delirium when giving midazolam compared to propofol, hypoglycemia when giving a continuous insulin drip in high doses and giving a lower amount of calories to a patient who will receive TPN without lipids.

There are many studies that examined the administration of vitamin C to patients in intensive care, especially patients with sepsis, with varied but inconclusive results. A recently published meta-analysis found a reduction in mortality among critical intensive care patients treated with intravenous vitamin C, especially in the subgroup of critically ill patients with a high risk of in-hospital mortality. The drug was found to be safe for use among patients in intensive care. In these patients in the various studies, vitamin C treatment was given intravenously in different doses, with most patients receiving a dose of 6 grams per day for 3-5 days. In light of a trend about five years ago that showed an improvement in survival among septic patients in intensive care who were treated with intravenous vitamin C as monotherapy, or in combination with steroids and/or intravenous thiamine, also in the intensive care unit at our institution (as well as in other hospitals) we started giving this treatment, at the recommended dose of 6 grams per day for 3-5 days. Over time, new studies did not find clear benefits for this treatment, so we gradually stopped giving it. However, if indeed vitamin C can contribute to a significant decrease in TG levels in patients in intensive care, there may be a point in administering it to a group of patients with high TG levels, in order to reduce complications associated with a high TG level and/or treatment to reduce it.

ELIGIBILITY:
Inclusion Criteria: patients aged 18-99 who were admitted to the general intensive care unit from January 2017 to December 2023, and who were treated with intravenous vitamin C. The control group will include patients with the same characteristics who were not treated with vitamin C.

Exclusion criteria: patients who did not meet the above conditions or for whom data were missing.

-

-

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients aged 18-99 who were admitted to the general intensive care unit from January 2017 to December 2023, and who were treated with intravenous vitamin C. The control group will include patients with the same characteristics who were not treated with vitamin C.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin C administration and triglycerides level | 1 week from Vitamin C administration
  Changes in triglycerides level (mg/dl) after 3 days of vitamin C administration (6 gr/day IV )

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided